CLINICAL TRIAL: NCT05905770
Title: Do Serum Alemtuzumab Concentrations Predict Donor T Cell Chimerism After Non-Myeloablative Matched Sibling Donor Stem Cell Transplantation in Sickle Cell Disease Patients
Brief Title: Do Alemtuzumab Levels Predict T Cell Chimerism After MSD SCT for SCD?
Acronym: PREDICT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Erfan Nur, Prinicpal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: METC 2022_0189
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Allogeneic stem cell transplantation; Alemtuzumab
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Alemtuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood (serum)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sickle cell disease patients aged 16 years and older with an available matched sibling donor.: Alemtuzumab 1mg/kg/TBI 3Gy conditioning
  Interventions: Drug: Alemtuzumab Injection [Campath]

INTERVENTIONS:
Drug: Alemtuzumab Injection [Campath] — Alemtuzumab 1mg/kg

SUMMARY:
Rationale: Non-myeloablative allogeneic stem cell transplantation (SCT) has become a feasible curative treatment option for sickle cell disease (SCD) patients with an available matched sibling donor. Chemotherapy free conditioning with alemtuzumab and 3 Gy total body irradiation (TBI) is increasingly being used as preferred conditioning scheme for these patients. This regimen typically results in mixed donor chimerism and has only few toxic effects. However, the risk of graft failure (rejection) is still significant, with an occurrence of 13% in the latest series. Levels of T cell chimerism are crucial for the success of this kind of transplantation. A donor T cell level of at least 50% at 1-year post-transplantation seems to be sufficient to allow the discontinuation of immunosuppressive medication without risk of graft rejection. Low levels of alemtuzumab prior to or shortly after SCT are thought to facilitate rejection of the donor graft. Recently, a positive correlation between alemtuzumab levels on day+14 was found with levels of T cell chimerism +2 and +4 months post-transplantation in adult SCD patients receiving matched sibling donor SCT. However, in this study alemtuzumab levels prior to the infusion of hematopoietic stem cells and beyond day +28 post-transplantation were not measured. Furthermore, the alemtuzumab levels were measured in 2 patient groups undergoing two different conditioning regimens.

Here, the investigators aim to thoroughly investigate the correlation of alemtuzumab levels and T cell chimerism. This will be the first study involving SCD patients receiving matched sibling donor SCT with alemtuzumab/TBI conditioning that includes alemtuzumab level measurements before the infusion of hematopoietic stem cells and beyond 1-month post-transplantation. Findings from this study will improve the insights into the etiology of graft failure in these patients and might ultimately lead to a more personalized approach in dosing alemtuzumab in order to achieve a more robust and stable engraftment of donor hematopoietic stem cells.

Objectives: To investigate whether serum alemtuzumab concentrations are predictive of the robustness of engraftment in SCD patients undergoing a matched sibling donor transplantation with alemtuzumab/TBI conditioning resulting in mixed chimerism.

Study design: Prospective observational laboratory study. Serum alemtuzumab concentration will be measured at various time points before and after stem cell infusion (days -3, 0, +7, +14, +28, +60).

Study population: Adult SCD patients that are planned for a matched sibling donor transplantation with alemtuzumab/TBI conditioning at the Amsterdam UMC.

Main study parameters/endpoints: The correlation between serum alemtuzumab concentration and levels of donor chimerism. Secondary endpoints: correlation between serum alemtuzumab levels and patients with and without successful engraftment. Correlation of serum alemtuzumab levels and the dosing of alemtuzumab in mg/kg, number of patient lymphocyte count and total number of infused enucleated donor-derived cells.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years and older
* High performance liquid chromatography (HPLC) confirmed diagnoses of SCD (all genotypes)
* Planned for a non-myeloablative matched sibling donor SCT with alemtuzumab/TBI at the Amsterdam UMC
* Willing and able to provide written informed consent

Exclusion Criteria:

* No specific exclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult SCD patients that are planned for a matched sibling donor transplantation with alemtuzumab/TBI conditioning at the Amsterdam UMC.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The correlation between serum alemtuzumab concentration and donor T cell chimerism. | +1 year post-transplantation

SECONDARY OUTCOMES:
o The differences in serum alemtuzumab concentration at the various time points (T1-T7) between patients with and without successful engraftment. Successful engraftment is defined as donor T cell chimerism >50% at 1-year post-transplantation. | +1 year post-transplantation
o The correlation between the dosing of alemtuzumab in mg/kg, the number of patient lymphocytes and alemtuzumab levels at the various time points (T1-T7). | +1 year post-transplantation
o The correlation between total number of infused enucleated donor-derived cells and the amount of decrease of alemtuzumab levels before and after stem cell infusion (T2 and T3). | +1 year post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Erfan Nur, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam Medical Centre, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided